CLINICAL TRIAL: NCT06982963
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate the Efficacy and Safety of FB102 in Adult Participants With Celiac Disease on a Gluten Free Diet
Brief Title: Randomized, Double Blind, Placebo-controlled Phase 2 Study in Adults With Celiac Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Forte Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB102-301
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): FB102
  Interventions: Biological: FB102
- B (Experimental): FB102
  Interventions: Biological: FB102
- C (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: FB102 — FB102 (10 mg/kg induction doses and 3 mg/kg or 5 mg/kg maintenance doses) or placebo arms in a 2:2:1 ratio.
  Arms: A; B
Other: Placebo — Placebo
  Arms: C

SUMMARY:
This study is a randomized, double-blind, placebo controlled clinical study to assess the efficacy, safety, pharmacokinetics (PK) and pharmacodynamics (PD) of FB102 in adult participants with well controlled (on a strict GFD) CeD following an oral gluten challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 70 years at Screening.
2. Has documented diagnosis of CeD confirmed by intestinal biopsy and positive celiac serology at least 12 months prior to Screening (intestinal biopsy and serology do not have to be performed concurrently).
3. Body mass index (BMI) between 16.0 and 40.0 kg/m2, inclusive.
4. Self-reported to be on a GFD for at least 12 months prior to Screening and must be willing to remain on a GFD for the duration of study participation, with the exception of the oral gluten challenge administered as a study procedure. Prior acute and resolved accidental exposures are not exclusionary.

Exclusion Criteria:

1. Uncontrolled CeD and/or active signs/symptoms of CeD, in the opinion of the Investigator.
2. History of or current neuropsychiatric manifestations specifically related to gluten exposure including ataxia, seizures, severe peripheral neuropathy, cognitive impairment, and depression.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the VCIEL | 78 Days
  Vh:Cd and IEL Composite Scale (VCIEL)

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: Undecided